CLINICAL TRIAL: NCT00351299
Title: Study of Dexmedetomidine as an Effective Sedative to Treat Acute ICU Delirium
Brief Title: Randomized Controlled Trial of Dexmedetomidine for the Treatment of Intensive Care Unit (ICU) Delirium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gerald L. Weinhouse, Staff Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-P-001786, BWH
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Delirium; Agitation
Keywords: Delirium; Agitation; Sedation; Dexmedetomidine; Surgical
MeSH Terms: conditions — Delirium; Psychomotor Agitation | interventions — Dexmedetomidine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion of dexmedetomidine (Experimental): infusion 0.3-0.7 dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Standard of Care (Other): Standard of care per treating physician preference
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine infusion titrated to effect
  Other Names: Precedex
  Arms: Infusion of dexmedetomidine
Other: Standard of Care — Standard of care per treating physician preference
  Arms: Standard of Care

SUMMARY:
The purpose of the research is to see if dexmedetomidine (a drug that has a calming effect - a sedative) is effective for the treatment of acute delirium

DETAILED DESCRIPTION:
Delirium is a mental disturbance that causes people to be confused and restless for a period of time. We will compare dexmedetomidine to the traditional therapy for treatment of acute delirium. Dexmedetomidine does not affect breathing. The traditional drugs might make one sleepy and may slow down breathing. The traditional therapy in this institution for acute delirium is _the use of Haloperidol, and/or benzodiazepines. Haloperidol is an antipsychotic drug that has calming effect. Benzodiazepines are sedatives with calming effect.Dexmedetomidine is approved by the Food and drug Administration (FDA) to sedate patients on a breathing machine for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to our surgical ICU who do not have any exclusion criteria
* Eligibility for treatment- Development of delirium as defined

Exclusion Criteria:

* Acute MI (myocardial infarction),
* Trauma <24 hours,
* Head injury,
* Multiple organ failure,
* EF (ejection fraction) < 30%,
* History of hypersensitivity to alpha2 agonist,
* History of seizures, MAP (mean arterial pressure) <60 mm of Hg,
* Dysrhythmias a/with bradycardia (HR (heart rate) <50),
* Need for vasopressors,
* Acute renal failure with a need for dialysis/CVVH (Continuous Veno-Venous Hemofiltration) or liver disease.
* Women of child bearing age who do not have a documented negative pregnancy test and/or who do not actively use contraception. (Documented negative pregnancy test will be a urine pregnancy test obtained on this admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald L Weinhouse, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to ICU from 2005-2008
Pre-assignment Details: Patients enrolled and randomized upon admission to ICU but treated with dexmedetomidine or standard of caremodalities only if they developed delirium.
Groups:
- Infusion of Dexmedetomidine: infusion 0.2-0.7 dexmedetomidine
  Dexmedetomidine: dexmedetomidine infusion titrated to effect
Period: Overall Study
Arm/Group | Infusion of Dexmedetomidine | Standard of Care
Started | 25 | 28
Completed | 25 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infusion of Dexmedetomidine | Standard of Care | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.00 (10.36) | 63.93 (11.55) | 63.96 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 17 | 21 | 38
Region of Enrollment [Number; unit: participants]
  United States | 25 | 28 | 53

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Delirium
Description: Resolution of delirium as defined by 2 consecutive negative CAM-ICU assessments.
  The Confusion Assessment Method for the ICU (CAM-ICU). The CAM-ICU assesses the four features of delirium: feature 1 is an acute change in mental status or a fluctuating mental status, feature 2 is inattention, feature 3 is altered level of consciousness, and feature 4 is disorganized thinking.
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care: Standard of Care Per treating attending physician preference
Arm/Group | Infusion of Dexmedetomidine | Standard of Care
Number analyzed (Participants) | 25 | 28
Participants | 21 | 14

2. Secondary Outcome: Length of Ventilator Support
Description: Number of days on mechanical ventilation
Time Frame: Patients will remain in the study for up to 7 days after development of delirium or discharge from ICU whichever is earlier, up to study end
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Infusion of Dexmedetomidine | Standard of Care
Number analyzed (Participants) | 25 | 28
days | 1 [0 to 4] | 2 [0.50 to 15.50]

3. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Description: Number of days intensive care unit (ICU) stay
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Standard of Care: Standard of Care Per attending physician preference
Arm/Group | Infusion of Dexmedetomidine | Standard of Care
Number analyzed (Participants) | 25 | 28
days | 7 [5 to 11] | 7.5 [5 to 19]

4. Secondary Outcome: Ease of Management for the Nursing Staff
Description: Subjective measure rating 3 categories for ease of management:
  1. Mostly easy
  2. Easy to manage 75% of the time
  3. Not easy to manage
Time Frame: Up to initial 48 hours
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care: Standard of care per attending physician's preference
Arm/Group | Infusion of Dexmedetomidine | Standard of Care
Number analyzed (Participants) | 25 | 28
Participants
  Mostly easy | 16 | 7
  Easy to manage 75% of the time | 4 | 2
  Not easy to manage | 5 | 19

5. Secondary Outcome: In-hospital Mortality
Description: Did patient die while in the hospital? (Yes/No)
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care: Standard of Care Per treating physician's preference
Arm/Group | Infusion of Dexmedetomidine | Standard of Care
Number analyzed (Participants) | 25 | 28
Participants
  Yes, died | 1 | 5
  No, did not die | 24 | 23

ADVERSE EVENTS:
Arm/Group | Infusion of Dexmedetomidine | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/28
Other Adverse Events (participants affected / at risk) | 0/25 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes